CLINICAL TRIAL: NCT06011317
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of EDG-7500 in Healthy Adults
Brief Title: A Study of EDG-7500 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Edgewise Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: EDG-7500-101
Record Dates: First submitted 2023-08-13; First posted 2023-08-25 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: Healthy Volunteer (Ages ≥ 18 to < 60 years) Single Ascending Dose (Experimental): Single oral ascending dose in healthy volunteers ages ≥ 18 to < 60 years
  Interventions: Drug: EDG-7500; Drug: Placebo
- Part B: Healthy Volunteer (Ages ≥ 18 to < 60 years) Multiple Ascending Doses (Experimental): Multiple oral ascending doses in healthy volunteers ages ≥ 18 to < 60 years
  Interventions: Drug: EDG-7500; Drug: Placebo
- Part D: Healthy Volunteer Food Effect and Relative Bioavailability (Experimental): Crossover food effect (fed versus fasted) single oral dose in healthy volunteers and relative bioavailability of liquid versus solid formulation
  Interventions: Drug: EDG-7500

INTERVENTIONS:
Drug: EDG-7500 — EDG-7500 is administered orally once daily
Drug: Placebo — Placebo is administered orally once daily
  Arms: Part A: Healthy Volunteer (Ages ≥ 18 to < 60 years) Single Ascending Dose; Part B: Healthy Volunteer (Ages ≥ 18 to < 60 years) Multiple Ascending Doses

SUMMARY:
The purposes of this Phase 1 study of EDG-7500 are to:

1. Learn about the safety of EDG-7500 after a single and multiple doses in healthy adults
2. Learn about how EDG-7500 is tolerated after a single and multiples doses in healthy adults
3. Evaluate the amount of EDG-7500 is in the blood and urine after single and multiple doses in healthy adults
4. Evaluate the effect of a meal on the amount of EDG-7500 that is in the blood in healthy adults
5. Evaluate whether the amount of EDG-7500 in the blood is similar for the suspension and tablet forms of EDG-7500 in healthy adults

Participants will receive a single or multiple doses of EDG-7500 or a placebo by mouth.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give informed consent and follow all study procedures and requirements.
2. Healthy male or nonpregnant female, ages ≥ 18 to < 60 years.
3. Body mass index (BMI) ≥ 18 to < 35 kg/m2; weight ≥ 55 kg at Screening.
4. Absence of important health problems and essentially normal physical examination, normal laboratory screening tests, and normal electrocardiogram (ECG) with QTcF ≤ 450 ms.

Exclusion Criteria:

1. Evidence of clinically significant abnormalities or disease.
2. Unless permitted by protocol, use of any prescription medication ≤ 4 weeks or investigational medication ≤ 12 weeks or ≤ 5 half-lives (whichever is longer) of dosing. Use of any non-prescription medication or herbal/nutritional supplement ≤ 5 days prior to dosing.
3. Donation or loss of > 1 unit (450 mL) of blood ≤ 1 month prior to dosing.
4. Females: nursing, lactating, or pregnant.
5. Females: breast implants.
6. Use of nicotine-containing products in the last 6 months prior to dosing.
7. History of substance abuse or dependency or history of recreational drug use. Alcohol consumption > 14 drinks per week for males (7 for females). Positive screen for drugs of abuse or alcohol or cotinine test at Screening or Admission.

Additional protocol defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Safety: incidence of treatment-emergent adverse events | Up to 25 days of monitoring
  To assess the safety and tolerability of EDG-7500 when administered as single and multiple doses

SECONDARY OUTCOMES:
Determination of pharmacokinetics parameters as measured by Tmax | Up to 25 days of monitoring
  Time to maximum concentration (Tmax)
Determination of pharmacokinetic parameters as measured by Cmax | Up to 25 days of monitoring
  Maximum observed concentration (Cmax)
Determination of pharmacokinetic parameters as measured by AUC | Up to 25 days of monitoring
  Area under the concentration-time curve (AUC)
Determination of pharmacokinetic parameters as measured by t1/2 | Up to 25 days of monitoring
  Terminal half-life (t1/2)
Determination of renal clearance as measured by CLr | Up to 25 days of monitoring
  Renal clearance (CLr)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Edgewise Therapeutics, Inc.
Locations (2):
- United States (2):
  - Celerion, Tempe, Arizona
  - Celerion, Lincoln, Nebraska

IPD SHARING:
Plan to Share IPD: No